CLINICAL TRIAL: NCT03701867
Title: A Pilot Study to Explore Muscle Energy Metabolism and Metabolic Flexibility in Older Men and Women
Brief Title: Muscle Energy Metabolism and Metabolic Flexibility in Older Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BL39
Record Dates: First submitted 2018-09-21; First posted 2018-10-10 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Energy Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metabolic Flexibility Tests Group (Experimental)
  Interventions: Other: Metabolic Flexibility Tests

INTERVENTIONS:
Other: Metabolic Flexibility Tests — Energy Metabolism, Oxygenation, Body Composition, Blood Samples

SUMMARY:
This study will explore differences in energy metabolism and metabolic flexibility under various conditions in older men and women.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >20.0 and <39.0 kg/m2
* Ambulatory (may use assistance device e.g., cane, walker)
* Not a current smoker (within past 10 years)
* Low or moderate risk based on the responses from the AHA/ACSM Health/Fitness Facility Preparticipation Screening Questionnaire
* Normal muscle mass and strength/performance or sarcopenia included in low muscle mass and low grip strength
* If on thyroid medication or hormone replacement therapy, has been on a constant dosage for at least 2 months prior to Screening Visit
* Willingness to follow protocol as described
* Voluntarily signed and dated an informed consent form (ICF), approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB) prior to any participation in the study

Exclusion Criteria:

* Active/treated disease, under the care of a physician, for the following: metabolic/endocrine (diabetes), hepatic, or renal disease, myocardial infarction, peripheral vascular disease, respiratory or neuromuscular disease
* Participates in a resistance exercise program
* Poor appetite with recent unexplained weight loss over the past 6 months
* Current infection (requiring medication or which might be expected to require hospitalization); has had inpatient surgery, or corticosteroid treatment (excluding topical creams) in the last 3 months or antibiotics in the last 3 weeks.
* Active malignancy, excluding carcinoma in-situ of the cervix, cutaneous malignancies (basal cell carcinoma, squamous cell carcinoma, except melanoma)
* Chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis A, B or C, or HIV
* Taking medications/dietary supplements or substances that could profoundly modulate metabolism in the opinion of the principal investigator or study physician, Exceptions for multi-vitamin/mineral supplement, topical or optical steroids and short-term use (less than two weeks) of dexamethasone
* Allergy or intolerance to any foods
* History of gastrointestinal disease, or surgeries, gastroparesis, or taking medications that are known in the opinion of the PI or study physician to interfere with consumption/digestion/absorption of nutrients
* Eating disorder, severe dementia or delirium, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with compliance with study protocol procedures in the opinion of the principal investigator or study physician
* Participant in a concomitant AN trial or trial of a non-registered drug (or is within the 30 day follow-up period for such a trial) or that otherwise conflicts with this study unless otherwise approved

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Respiratory Quotient | Baseline to 270 minutes
  Ratio of macronutrient oxidation

SECONDARY OUTCOMES:
Blood Biochemistries - Glucose | Baseline to 270 minutes
  Venous blood sample
Blood Biochemistries - Insulin | Baseline to 270 minutes
  Venous blood sample
Blood Biochemistries - Amino Acids | Baseline to 270 minutes
  Venous blood sample
Blood Biochemistries - Fatty Acids | Baseline to 270 minutes
  Venous blood sample
Muscle Oxygenation | Baseline to 270 minutes
  Near Infrared Spectroscopy
Muscle Fatigue | Baseline to 270 minutes
  Electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Vikkie Mustad, PhD, Study Chair — Abbott Nutrition
Locations (1):
- University of Nebraska, Lincoln, Nebraska, United States

REFERENCES:
- [Derived] Shoemaker ME, Pereira SL, Mustad VA, Gillen ZM, McKay BD, Lopez-Pedrosa JM, Rueda R, Cramer JT. A pilot study evaluating differences in muscle tissue saturation and blood flow between older adults with and without sarcopenia. Front Endocrinol (Lausanne). 2025 Aug 13;16:1644712. doi: 10.3389/fendo.2025.1644712. eCollection 2025. PMID 41070343
- [Derived] Shoemaker ME, Pereira SL, Mustad VA, Gillen ZM, McKay BD, Lopez-Pedrosa JM, Rueda R, Cramer JT. Differences in muscle energy metabolism and metabolic flexibility between sarcopenic and nonsarcopenic older adults. J Cachexia Sarcopenia Muscle. 2022 Apr;13(2):1224-1237. doi: 10.1002/jcsm.12932. Epub 2022 Feb 17. PMID 35178889